CLINICAL TRIAL: NCT01168271
Title: Host and Parasite Factors That Influence Susceptibility to Malaria Infection and Disease During Pregnancy and Early Childhood in Ouelessebougou and Bamako, Mali
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910156; 10-I-N156
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-04-07

CONDITIONS: Malaria
Keywords: Observational; Newborns; Hospitalized; Febrile; Resistance; Natural History
MeSH Terms: conditions — Malaria; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Children Ages 0-3 years: Children aged 0-3 years in Ouelessebougou
- Febrile Hospitalized Children: Febrile hospitalized children aged 0-10 years in Ouelessebougou or the Pediatric service of Gabriel Toure Hospital in Bamako
- Later Childhood and Adolescence: Re-enrollees who were originally enrolled at birth and completed the Pregnant Women and Newborn Cohort
- Non-Hospitalized Children: Febrile non-hospitalized children aged 0-10 years in Ouelessebougou or the Pediatric service of Gabriel Toure Hospital in Bamako
- Pregnant Women + Newborns: Pregnant women presenting for antenatal consultations and delivery and their newborns

SUMMARY:
Malaria caused by Plasmodium falciparum continues to be a global problem with devastating consequences. A greater understanding of the immunologic and parasitologic factors associated with infection and disease is badly needed, and will accelerate the development of highly protective vaccines for both mothers and children. Pregnancy malaria is associated with low birth weight, maternal anemia, and gestational hypertension, and both inflammation and the fetal response to infection may contribute to these poor outcomes. Childhood malaria is a major cause of mortality, and we have found that risk of childhood malaria is related to in utero exposure to pregnancy malaria, as well as other host factors like iron status and constitutive cytokine levels. Pregnancy malaria is caused by a distinct parasite binding phenotype, and as our primary hypothesis in this study we speculate that severe childhood malaria parasites may also have distinct features. A longitudinal cohort study will be conducted in Ouelessebougou, Mali an area of intense seasonal transmission. Up to 2000 pregnant women and their infants and 2000 children ages 0 - 3 will be enrolled and followed to age 5 years, with clinical evaluation and periodic venous and peripheral blood samples obtained. In addition, 2000 febrile children up to age 10 years will be enrolled at the Ouelessebougou district health centers or the Gabriel Toure Pediatric Hospital in Bamako, Mali, with acute and convalescent samples being obtained and 500 pregnant women enrolled at the health centers and hospital in Ouelessebougou district or the Gabriel Toure Hospital in Bamako for a case-control study on pregnancy malaria and preeclampsia. Clinical, parasitologic and host response (including immunologic) endpoints will be analyzed using appropriate statistical methods, including possible confounders, to determine factors associated with infection and disease in pregnant woman and young children.

DETAILED DESCRIPTION:
Malaria caused by Plasmodium falciparum continues to be a global problem with devastating consequences. A greater understanding of the immunologic and parasitologic factors associated with infection and disease is badly needed; and will accelerate the development of highly protective vaccines for both mothers and children. Pregnancy malaria is associated with low birth weight, maternal anemia, and gestational hypertension, and both inflammation and the fetal response to infection may contribute to these poor outcomes. Childhood malaria is a major cause of mortality, and we have found that risk of childhood malaria is related to in utero exposure to pregnancy malaria, as well as other host factors like iron status and constitutive cytokine levels. Pregnancy malaria is caused by a distinct parasite binding phenotype, and as our primary hypothesis in this study we speculate that severe childhood malaria parasites may also have distinct features. A longitudinal cohort study will be conducted in Ouelessebougou, Mali, an area of intense seasonal transmission. Up to 2000 pregnant women and their infants and 2000 children ages 0-3 years will be enrolled and followed to age 5 years, with clinical evaluation and periodic venous and peripheral blood samples being obtained. In addition, up to 3000 febrile hospitalized and non-hospitalized children up to age 10 years will be enrolled at the Ouelessebougou district health centers or the Gabriel Toure Pediatric Hospital in Bamako, Mali, with acute and convalescent samples being obtained and 500 pregnant women enrolled at the health centers and hospital in Ouelessebougou district or the Gabriel Toure Hospital in Bamako for a case-control study on pregnancy malaria and preeclampsia. Up to 1000 children originally enrolled at birth and completed the "pregnant women and their newborns study" will be re-enrolled and followed-up for up to 10 years as they age from later childhood through adolescence to early adulthood. Clinical, parasitologic and host response (including immunologic) endpoints will be analyzed using appropriate statistical methods, including possible confounders, to determine factors associated with infection and disease in pregnant women and young children.

ELIGIBILITY:
* INCLUSION CRITERIA:

A study participant must satisfy the following criteria to be enrolled in this study:

1. Pregnant women aged 15-45 years and their newborn infants who are residents of the district of Ouelessebougou for at least one year at the time of enrollment; OR
2. Children who previously participated in the 1st cohort of "pregnant women and their newborn infants", OR
3. Children aged 3 years or less, who are residents of the district of Ouelessebougou for at least one year at the time of enrollment, OR
4. Febrile hospitalized children (aged 0-10 years), including those with positive and negative blood smears for P. falciparum in Ouelessebougou or the pediatric service of Gabriel Toure Hospital in Bamako. Febrile non-hospitalized children (aged 0-10 years) with non-severe malaria will be recruited at outpatient clinics in Ouelessebougou district health hospital and nearby facilities, with no chronic or serious illness.
5. Pregnant women aged 15-25 in Ouelessebougou district health centers or maternity unit of Gabriel Toure Hospital in Bamako and for a case-control study of pregnancy malaria and preeclampsia. Cases include women with signs/symptoms of preeclampsia. Control pregnant women without signs/symptoms of preeclampsia will be recruited sequentially after identification of individual cases, matched for parity, age (+/-2 years) and pregnancy trimester.
6. The study participant or parent/guardian understands the study and gives informed consent for participation of themselves and/or their child, and agrees to have samples stored.

EXCLUSION CRITERIA:

A participant will be excluded from the study if any one or more of the following criteria are met:

1. Chronic, debilitating illness, other than malaria, determined by history and physical examination of mother or study participant.
2. Conditions that in the judgment of the investigator could increase the risk to the volunteer.
3. History of previous participation in a malaria vaccine trial.

Ages: 1 Day to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women presenting for antenatal consultations and delivery and their newborns; children aged 0-3 years in Ouelessebougou and Febrile children ages 0-10 years hospitalized and non-hospitalized in Ouelessebougou or the Pediatric service of Gabriel Toure Hospital in Bamako; Re-enrollees who were originally enrolled at birth and completed the Pregnant Women and Newborn Cohort
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2010-08-30 (Actual)

PRIMARY OUTCOMES:
Maternal, placental, parasite and host associated with resistence to malaria infection and diseases in children | up to 5 years for infants and children
  To assess the relationship between malaria exposure during pregnancy and maternal and fetal outcomes; and to determine factors (maternal, placental, parasite, and host) associated with susceptibility or resistance to malaria infection and diseases in children

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Mali (2):
  - Gabriel Toure Hospital, Bamako
  - Ouelessebougou Clinical Research Center, Wolossébougou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried M, Nosten F, Brockman A, Brabin BJ, Duffy PE. Maternal antibodies block malaria. Nature. 1998 Oct 29;395(6705):851-2. doi: 10.1038/27570. No abstract available. PMID 9804416
- [Background] Ho M, Singh B, Looareesuwan S, Davis TM, Bunnag D, White NJ. Clinical correlates of in vitro Plasmodium falciparum cytoadherence. Infect Immun. 1991 Mar;59(3):873-8. doi: 10.1128/iai.59.3.873-878.1991. PMID 1997437
- [Background] Muehlenbachs A, Mutabingwa TK, Edmonds S, Fried M, Duffy PE. Hypertension and maternal-fetal conflict during placental malaria. PLoS Med. 2006 Nov;3(11):e446. doi: 10.1371/journal.pmed.0030446. PMID 17105340
- [Derived] Doritchamou JYA, Renn JP, Jenkins B, Mahamar A, Dicko A, Fried M, Duffy PE. A single full-length VAR2CSA ectodomain variant purifies broadly neutralizing antibodies against placental malaria isolates. Elife. 2022 Feb 1;11:e76264. doi: 10.7554/eLife.76264. PMID 35103596
- [Derived] Mahamar A, Gonzales Hurtado PA, Morrison R, Boone R, Attaher O, Diarra BS, Gaoussou S, Issiaka D, Dicko A, Duffy PE, Fried M. Plasma biomarkers of hemoglobin loss in Plasmodium falciparum-infected children identified by quantitative proteomics. Blood. 2022 Apr 14;139(15):2361-2376. doi: 10.1182/blood.2021014045. PMID 34871370
- [Derived] Mahamar A, Andemel N, Swihart B, Sidibe Y, Gaoussou S, Barry A, Traore M, Attaher O, Dembele AB, Diarra BS, Keita S, Dicko A, Duffy PE, Fried M. Malaria Infection Is Common and Associated With Perinatal Mortality and Preterm Delivery Despite Widespread Use of Chemoprevention in Mali: An Observational Study 2010 to 2014. Clin Infect Dis. 2021 Oct 20;73(8):1355-1361. doi: 10.1093/cid/ciab301. PMID 33846719
- [Derived] Fried M, Kurtis JD, Swihart B, Pond-Tor S, Barry A, Sidibe Y, Gaoussou S, Traore M, Keita S, Mahamar A, Attaher O, Dembele AB, Cisse KB, Diarra BS, Kanoute MB, Dicko A, Duffy PE. Systemic Inflammatory Response to Malaria During Pregnancy Is Associated With Pregnancy Loss and Preterm Delivery. Clin Infect Dis. 2017 Oct 30;65(10):1729-1735. doi: 10.1093/cid/cix623. PMID 29020221